CLINICAL TRIAL: NCT04906655
Title: An Open-label Study to Evaluate the Efficacy and Safety of Different Methods of Application of Glycopyrronium Cloth, 2.4% in Patients With Palmar Hyperhidrosis
Brief Title: An Open Label Study for Palmar Hyperhydrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pariser, Robert J., M.D. (Other)
Collaborators: Virginia Clinical Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PQB-001
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Palmar Hyperhidrosis; Hyperhidrosis; Sweat Gland Diseases; Skin Diseases
Keywords: QBREXZA; glycopyrronium
MeSH Terms: conditions — Hyperhidrosis; Sweat Gland Diseases; Skin Diseases | interventions — Glycopyrrolate; glycopyrronium tosylate

STUDY DESIGN:
Intervention Model Description: The study is open label, and treatment groups are assigned by Cohorts starting with A, then B, then C, then D. The method of treatment will be filled on a first come, first served basis. Movement from one cohort to the next will be determined by the medical monitor after evaluation of the safety and efficacy data that is available after each cohort is filled. There may be a very brief enrollment (baseline) pause for this to occur.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort A glycopyrronium 30 minutes cotton gloves (Experimental): Study drug should be applied to clean, dry skin. A single cloth will be used to apply study drug to both hands once daily, at bedtime. The subject will be instructed to apply the study drug as follows:
  30 minutes residence time in cotton gloves
  1. Complete daily diary.
  2. Remove all jewelry.
  3. Tear open the top of the pouch at the notch.
  4. Wash hands thoroughly with warm water, and dry them.
  5. Remove the wipe from the pouch and unfold the wipe.
  6. Wipe both hands with the wipe continuously until the wipe is dry (up to 3 minutes).
  7. Return the wipe to the pouch and put it back in the box.
  8. Carefully put cotton gloves on both hands.
  9. Set timer for 30 minutes.
  10. After 30 minutes, remove gloves and throw them away. Immediately wash hands thoroughly with warm water and soap, and dry them.
  Interventions: Drug: Glycopyrronium 2.4 % Medicated Cloth
- Cohort B glycopyrronium 30 minutes under occlusion (Experimental): Study drug should be applied to clean, dry skin. A single cloth will be used to apply study drug to both hands once daily, at bedtime. The subject will be instructed to apply the study drug as follows:
  30 minutes residence time under occlusion
  1. Complete daily diary.
  2. Remove all jewelry.
  3. Tear open the top of the pouch at the notch.
  4. Wash hands thoroughly with warm water, and dry them.
  5. Remove the wipe from the pouch and unfold the wipe.
  6. Wipe both hands with the wipe continuously until the wipe is dry (up to 3 minutes).
  7. Return the wipe to the pouch and put it back in the box.
  8. Carefully put gloves on both hands.
  9. Set timer for 30 minutes.
  10. After 30 minutes, remove gloves and throw them away. Immediately wash hands thoroughly with warm water and soap, and dry them.
  Interventions: Drug: Glycopyrronium 2.4 % Medicated Cloth
- Cohort C glycopyrronium overnight in cotton gloves (Experimental): Study drug should be applied to clean, dry skin. A single cloth will be used to apply study drug to both hands once daily, at bedtime. The subject will be instructed to apply the study drug as follows:
  Overnight in cotton gloves
  1. Complete daily diary
  2. Remove all jewelry.
  3. Tear open the top of the pouch at the notch.
  4. Wash hands thoroughly with warm water, and dry them.
  5. Remove the wipe from the pouch and unfold the wipe.
  6. Wipe both hands with the wipe continuously until the wipe is dry (up to 3 minutes).
  7. Return the wipe to the pouch and put it back in the box.
  8. Carefully put on the cotton gloves on both hands and go to bed.
  9. In the morning, after at least 4 hours of wearing the gloves , remove the cotton gloves and throw them away.
  10. Immediately wash hands thoroughly with warm water and soap, and dry them.
  Interventions: Drug: Glycopyrronium 2.4 % Medicated Cloth
- Cohort D glycopyrronium overnight under occlusion (Experimental): Study drug should be applied to clean, dry skin. A single cloth will be used to apply study drug to both hands once daily, at bedtime. The subject will be instructed to apply the study drug as follows:
  Overnight under occlusion
  1. Complete daily diary
  2. Remove all jewelry.
  3. Tear open the top of the pouch at the notch.
  4. Wash hands thoroughly with warm water, and dry them.
  5. Remove the wipe from the pouch and unfold the wipe.
  6. Wipe both hands with the wipe continuously until the wipe is dry (up to 3 minutes).
  7. Return the wipe to the pouch and put it back in the box.
  8. Carefully put on the occlusive gloves and go to bed.
  9. In the morning, after at least 4 hours of wearing the gloves, remove the occlusive gloves and throw them away.
  10. Immediately wash hands thoroughly with warm water and soap, and dry them.
  Interventions: Drug: Glycopyrronium 2.4 % Medicated Cloth

INTERVENTIONS:
Drug: Glycopyrronium 2.4 % Medicated Cloth — The investigational product (glycopyrronium cloth, 2.4%) is a pre-moistened, medicated cloth towelette that comes in individually wrapped packets. Subjects will receive marketed Qbrexza, one box, containing 30 pouches.
  Other Names: Qbrexza

SUMMARY:
The purpose of this open-label study is to evaluate the efficacy and safety of different methods of application of glycopyrronium cloth, 2.4% in patients with palmar hyperhidrosis

DETAILED DESCRIPTION:
This study will assess glycopyrronium cloth, 2.4% in patients with primary palmar hyperhidrosis and compare the efficacy and safety of various application methods in order to determine an optimal method for use in palmar hyperhidrosis. The study will assess four application methods (treatment groups). Data from these cohorts will be reviewed on a continuous basis, and the protocol may be amended to add one or more treatment groups if required to determine the optional conditions of drug application.

This study is open label and unblinded. The treatment groups will be enrolled in cohorts, with each cohort being filled before moving on to the next. Cohort A will be enrolled first, followed by B, C, and D. Each cohort will have 30 subjects. If there are multiple AEs of special interest, the medical monitor may stop enrollment of one or more cohorts or may prematurely terminate a cohort(s).

All visits for this study will be conducted virtually, using HIPAA compliant video conferencing technology. Investigational product (IP) will be shipped overnight to subjects that are deemed eligible for participation.

All subjects will sign an informed e-consent and undergo screening for study eligibility. Key criteria for entry are: primary palmar hyperhidrosis for at least 6 months, an average hand sweat severity score of ≥4 (NRS 0-10 pts) during the screening period. Exclusion criteria includes pregnancy or lactation, secondary hyperhidrosis, prior sympathectomy, open wounds or infection on the hands, and concomitant use of iontophoresis, botulinum toxin, experimental therapy, or unstable doses of anticholinergic medications. Subjects will only be allowed to enroll into one cohort.

Approximately 120 eligible subjects, ≥9 years of age will be enrolled to one of four treatment groups at the Baseline visit.

Cohort Table 1: Treatment Groups A 30 minutes residence time in cotton gloves n=30 B 30 minutes residence time under occlusion n=30 C Overnight in cotton gloves n=30 D Overnight under occlusion n=30

Subjects will be instructed on the application method and will apply study drug at home once each evening before going to bed for 28 days (+/- 2 days). Subjects will complete virtual visits to check for adverse events (AEs) and study drug compliance at Week 1, Week 2, and Week 4. Subjects will exit the study at the Week 4 visit.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for study participation.

1. Subjects must provide fully executed informed e-consent and e-assent (if applicable) prior to any study procedures.
2. Age ≥ 9 years.
3. Willing to comply with the protocol, including completion of designated virtual study visits and prescribed study treatment regimens.
4. Subjects must have access to and the ability and willingness to use their own smart device (e.g., phone, computer, tablet). Subjects must have reliable internet access and video capabilities to conduct virtual visits, e-consent, and ePROs. Subjects must have an active email address that is password protected. Their password must remain confidential throughout the study.
5. Subjects must have a street address to which study drug can be delivered and received in a timely manner. (PO Boxes will not be allowed.)
6. Male or non-lactating and non-pregnant females (documentation of a negative urine pregnancy test done by the subject must be done prior to sending study drug.)
7. Primary palmar hyperhidrosis for at least 6 months.
8. Average sweat severity score of ≥4 at the end of screening. Subjects must complete the diary at least 4 times out of 7 days prior to baseline.
9. Females of childbearing potential must be willing to use an acceptable method of birth control during study participation and for 30 days after the last study drug application. Females are considered to be of childbearing potential unless surgically sterilized (hysterectomy, bilateral oophorectomy, tubal ligation), have been diagnosed as infertile, have same gender sex partner, or are postmenopausal for at least 1 year. Acceptable methods of contraception include: abstinence, oral contraceptives, contraceptive patches/implants, injectable contraceptives, double barrier methods (e.g., condom and spermicide), or an intra-uterine device (IUD). Birth control method must have been stable/unchanged for 12 weeks prior to Baseline and must remain unchanged during study participation and for 30 days after the last study drug application.
10. Males must either have been vasectomized or agree to use an acceptable method of birth control with female partners during study participation and for 30 days after the last study drug application.
11. Subjects must agree not to donate eggs or sperm (as applicable) during the trial.

    -

Exclusion Criteria:

Subjects meeting any of the following criteria are not eligible for study participation.

1. Prior surgical procedure for hyperhidrosis.
2. Iontophoresis for the palms within 4 weeks of Baseline.
3. Treatment with botulinum toxin (e.g., Botox®) for palmar hyperhidrosis within 1 year of Baseline. (Note: treatment with botulinum toxin in other areas is not exclusionary.)
4. Subjects who are actively participating in an experimental therapy study or who received experimental therapy within 30 days of 5 half-lives (whichever is longer) of the Baseline Visit.
5. For subjects that are taking concomitant medications that may have an effect on sweating (i.e., psychotherapeutic medications, centrally acting alpha-2 adrenergic agonists (e.g., clonidine, guanabenz, methyl dopa), or beta blockers, the dose must be stable, in the opinion of the investigator, for two months prior to Baseline. There should be no expected medication changes over the course of the study unless deemed to be medically necessary. (Note: inhaled anticholinergic drugs or beta agonists are allowed.)
6. Intravenous (IV), oral, or topically glycopyrrolate treatment of any systemic treatment with an anticholinergic medication, such as atropine, belladonna, scopolamine, clindinium, or hyoscyamine within 4 weeks prior to Screening.
7. Current pregnancy or lactation per patient report.
8. Open wounds or inflammatory lesions on the hands, or any condition that may alter the barrier function of the skin on the hands.
9. Secondary palmar hyperhidrosis or presence of a condition that may cause secondary hyperhidrosis (e.g., lymphoma, malaria, severe anxiety not controlled by medication, carcinoid syndrome, substance abuse, hyperthyroidism).
10. Known history of Sjögren's syndrome or Sicca syndrome.
11. History of glaucoma, inflammatory bowel disease, toxic megacolon, active febrile illness, paralytic ileus, unstable cardiovascular status in acute hemorrhage, severe ulcerative colitis, toxic megacolon complicating ulcerative colitis or myasthenia gravis.
12. Men with a history of urinary retention requiring catherization due to prostatic hypertrophy or severe obstructive symptoms of prostatic hypertrophy.
13. History of ventricular arrhythmias, atrial fibrillation, atrial flutter.
14. Subjects with known medical procedures or surgeries that are scheduled to occur during the study.
15. Subjects who are a poor medical risk because of other systemic diseases or active, uncontrolled infections, or any other condition, which (in the judgement of the investigator) would put the subjects at unacceptable risk for participation in the study.

    -

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Mean change of the average hand sweating score (Daily Diary Question 1) from the week of Screen-Baseline to the final week of study treatment. | From the week of Screen-Baseline (7 days prior to the end of the screening visit) to the final week of study treatment (week 4).
  The hand sweat severity (HSS) item is a patient reported outcome, collected nightly, and is designed to measure the severity of palmar hyperhidrosis.
Proportion of subjects who have a >2 grade improvement in HDSS from baseline to week 4. | From Baseline to week 4.
  Hyperhidrosis Disease Severity Scale (HDSS) is a disease specific diagnostic tool that provides a qualitative measure of the severity of the subjects' condition based on how it affects daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: David M Pariser, MD, Principal Investigator — Virginia Clinical Research, Inc.
Locations (1):
- Virginia Clinical Research, Inc., Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No